CLINICAL TRIAL: NCT01289366
Title: Endocytoscopy for in Vivo Determination of Mucosal Inflammatory Cells and Intestinal Disease Activity in Patients With Inflammatory Bowel Disease
Brief Title: Endocytoscopy for in Vivo Determination of Mucosal Inflammatory Cells and Intestinal Disease Activity in Inflammatory Bowel Disease (IBD)
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Markus F. Neurath, M.D., Ph.D., University of Erlangen-Nuremberg
Other Study IDs: HN-0006; Ecy1
Record Dates: First submitted 2011-02-02; First posted 2011-02-03 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Crohn´s Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with IBD
  Interventions: Device: Endocytoscopy

INTERVENTIONS:
Device: Endocytoscopy — Patients with Crohn's disease and ulcerative colitis who underwent colonoscopy are prospectively included in this study. Methylene blue or toluidine blue is topically applied to enable EC (XEC-120-U, Olympus, Tokyo, Japan). Data are digitally saved and analyzed independently from each other by two gastroenterologists and one pathologist who are blinded to clinical and endoscopic data.

SUMMARY:
Precise activity assessment of inflammatory bowel disease (IBD) is essential to determine the extent and severity of the disease for further specific therapy. Nevertheless, despite ongoing developments in the field of gastrointestinal endoscopy, the final diagnosis still relies on the interpretation of histopathological features of intestinal biopsies taken during the endoscopic examination. Recently, endocytoscopy (EC) was introduced as a new endoscopic imaging modality, enabling microscopic imaging within the mucosal layer of the gut at a magnification level of up to 1400-fold.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age 18-85 years
* Ability of subjects to understand character and individual consequences of clinical trial
* Subjects undergoing colonoscopy
* Patients with known Crohn´s disease or ulcerative colitis

Exclusion Criteria:

* Inability to provide written informed consent
* Severe Coagulopathy (Prothrombin time < 50% of control, Partial thromboplastin time > 50 s)
* Impaired renal function (Creatinine > 1.2 mg/dl)
* Pregnancy or breast feeding
* Active gastrointestinal bleeding
* Known allergy to methylene blue or toluidine blue
* Residing in institutions (e.g. prison)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Crohn's disease and ulcerative colitis who underwent colonoscopy.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To investigate the potential of endocytoscopy for in vivo detection of mucosal inflammatory cells. | 40 patients

SECONDARY OUTCOMES:
To evaluate the potential of endocytoscopy for the determination of intestinal inflammatory activity in patients with quiescent IBD and to compare endocytoscopy results with the results of standard histopathology | 40 patients

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Neumann, M.D., Ph.D., Principal Investigator — University of Erlangen-Nürnberg
Locations (1):
- University of Erlangen-Nuremberg, Erlangen, Bavaria, Germany

REFERENCES:
- [Derived] Neumann H, Vieth M, Neurath MF, Atreya R. Endocytoscopy allows accurate in vivo differentiation of mucosal inflammatory cells in IBD: a pilot study. Inflamm Bowel Dis. 2013 Feb;19(2):356-62. doi: 10.1002/ibd.23025. PMID 22644957